CLINICAL TRIAL: NCT03389165
Title: The Effect of a Wearable Hip Assist Robot on Cardiopulmonary Metabolic Efficiency During Stair Ascent in Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-08-028
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Gait, Unsteady; Health Behavior
Keywords: Wearable hip assist robot; Elderly adult; Metabolic energy expenditure; Stair ascent
MeSH Terms: conditions — Gait Disorders, Neurologic; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly adults (Experimental): Stair climbing with and without a wearable hip assist robot
  Interventions: Device: Wearable hip assist robot

INTERVENTIONS:
Device: Wearable hip assist robot — All participants climbed stairs from the first basement level to the fourth floor of the Proton Therapy Center, Samsung Medical Center, Korea with and without a wearable hip assist robot. During climbing stairs, the metabolic energy expenditure of all participants was measured using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy).

SUMMARY:
The aim of this study was to identify the assistance effect of the new wearable hip assist robot, gait enhancing mechatronic system (GEMS) developed by Samsung Advanced Institute of Technology (Samsung Electronics Co, Ltd., Korea) during stair ascent by comparing the energy expenditure of elderly adults with and without the GEMS.

DETAILED DESCRIPTION:
Primary objective of this study is to demonstrate the effect of a wearable hip assist robot on cardiopulmonary metabolic efficiency during stair ascent in elderly adults.

Fifteen elderly adults participated in this study. The stair ascent trials were designed to climb stairs from the first basement level to the fourth floor of the Proton Therapy Center, Samsung Medical Center, Korea. The metabolic energy expenditure was measured using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy) while participants performed randomly assigned two different conditions consecutively:, free ascent without the GEMS (NoGEMS) or robot-assisted ascent with the GEMS (GEMS). Participants rested for 10 minutes between the two trial conditions.

ELIGIBILITY:
Inclusion Criteria:

* Elderly adults who absence of a history of musculoskeletal or central nervous system diseases
* High levels of physical performance (SPPB > 8)

Exclusion Criteria:

* Elderly adults who absence of the ability to walk independently due to visual field defects, fractures, or severe muscle weakness
* Severe dizziness that might lead to falls
* Cognitive disorders that might be difficult to understand accurately in this study

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Change on metabolic energy expenditure in GEMS condition compared with NoGEMS condition | 1 hour
  All participants stood in a comfortable position for 5 minutes to obtain baseline variables before stair ascent. Participants were then asked to climb stairs from the first basement level to the fourth floor of the Proton Therapy Center, Samsung Medical Center, Korea, in a step-over-step manner under two different conditions, GEMS and NoGEMS. The GEMS and NoGEMS conditions were conducted in a random order, and just before the second condition, participants stood for 2～3 minutes to obtain baseline variables once more.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DS, Lee HJ, Lee SH, Chang WH, Jang J, Choi BO, Ryu GH, Kim YH. A wearable hip-assist robot reduces the cardiopulmonary metabolic energy expenditure during stair ascent in elderly adults: a pilot cross-sectional study. BMC Geriatr. 2018 Sep 29;18(1):230. doi: 10.1186/s12877-018-0921-1. PMID 30268096